CLINICAL TRIAL: NCT07030374
Title: Effects of Conscious Connected Breathing Exercises on Sexual Function, Sleep and Mood in Women With Fibromyalgia
Brief Title: Effects of Conscious Connected Breathing Exercises on Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adana City Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gulsum Uysal, Ass. Professor Gulsum Uysal, Adana City Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 253/05.12.2024
Record Dates: First submitted 2025-06-05; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia Syndrome; Fibromyalgia Impact Questionnaire; Breathing Pattern Disorder; Female Sexual Dysfunction (FSD); Sleep; Anxiety State
MeSH Terms: conditions — Fibromyalgia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: intervention group (participating breathing sessions) and control group (not participating breathing sessions)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (breathing session) group (Active Comparator): conscious connected breathing exercises
  Interventions: Other: conscious connected breathing exercises
- control group (No Intervention): no breathing exercises

INTERVENTIONS:
Other: conscious connected breathing exercises — conscious connected mouth breathing session where the diaphragm is activated
  Arms: intervention (breathing session) group

SUMMARY:
Our aim in this study is to investigate the effects of conscious connected breathing exercises on sexual function, sleep, and mood in fibromyalgia patients. The investigators want to clearly show how breathing exercises affect sexual function, sleep, and mood in fibromyalgia patients by comparing the results from the control and study groups before and immediately after the sessions. By experiencing and learning breathing sessions, participants can do it on their own, wherever they want, without the need for a specific tool or examination, and change their lifestyle.

DETAILED DESCRIPTION:
Natural CCB sessions were conducted 3 times monthly (every Monday) for approximately 1.5 hours from 16:30 to 18:00 pm by qualified breathing coach (GU). Volunteer participants were recruited randomly. Initially, they were apprised of the study's objectives and methodologies. Secondly, a researcher (GYO) gathered sociodemographic data to ascertain admission criteria. Demographic information, including the duration of follow-up since the diagnosis of FMS, chronic disease history, medications utilized, age, body mass index, and marital status, will be solicited and documented. Participants completed the Fibromyalgia Impact Questionnaire (FIQ), Hospital Anxiety and Depression Scale (HADS), and Jenkins Sleep Rating Scale (JSS) and Female Sexual Function Index (FSFI). The assessments will be administered again to the same participants following three sessions. The results of the pre- and post-surveys will be compared. Statistical analyses were conducted to compare the scores before and after the breathing exercises and evaluate the differences between the groups (study and controls). The control group consists of women diagnosed with fibromyalgia who did not participate in breathing sessions.

ELIGIBILITY:
Inclusion Criteria:

* Female fibromyalgia patients who applied to the Adana City Training and Research Hospital for physical therapy and rehabilitation outpatient clinic
* Patients with stable period of the disease (fibromyalgia)

Exclusion Criteria:

* Individuals diagnosed with schizoaffective illness,
* Individuals utilizing antipsychotic medications,
* Pregnant participants,
* Participants who did not finish three sessions

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with Fibromyalgia Syndrome
Enrollment: 60 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | comparision of scales before and immediately breathing exercises among groups
  The assessments will be administered again to the same participants following three sessions. The results of the pre- and post-surveys will be compared. Statistical analyses were conducted to compare the scores before and immediately after the breathing exercises and evaluate the differences between the groups (study and controls). The control group consists of women diagnosed with fibromyalgia who did not participate in breathing sessions.FIQ is to assess the effects of fibromyalgia. The questionnaire comprises ten principal inquiries. The maximum attainable score is 100, signifying a more severe clinical condition as value rise.
Hospital Anxiety and Depression Scale (HADS) | comparision of scales before and immediately breathing exercises among groups
  The assessments will be administered again to the same participants following three sessions. The results of the pre- and post-surveys will be compared. Statistical analyses were conducted to compare the scores before and immediately after the breathing exercises and evaluate the differences between the groups (study and controls). The control group consists of women diagnosed with fibromyalgia who did not participate in breathing sessions. The HADS consists of two subscales that evaluate both anxiety and depression. The scale typically consists of 14 items, divided equally into seven questions for the anxiety subscale and seven for the depression subscale. Each question pertains to a distinct emotional condition and allows patients to assess the emotional states they have encountered during a specified timeframe (usually within the last week).
Jenkins Sleep Rating Scale (JSS) | comparision of scales before and immediately breathing exercises among groups
  The assessments will be administered again to the same participants following three sessions. The results of the pre- and post-surveys will be compared. Statistical analyses were conducted to compare the scores before and immediately after the breathing exercises and evaluate the differences between the groups (study and controls). The control group consists of women diagnosed with fibromyalgia who did not participate in breathing sessions. The Jenkins Sleep Rating Scale (JSS), a measurement instrument for evaluating sleep disturbances. The questionnaire assessed issues such as "difficulty falling asleep, waking up several times during the night, not being able to sleep without waking up during the night, feeling tired and exhausted after waking up during a normal sleep period."
Female Sexual Function Index (FSFI) | comparision of scales before and immediately breathing exercises among groups
  The assessments will be administered again to the same participants following three sessions. The results of the pre- and post-surveys will be compared. Statistical analyses were conducted to compare the scores before and immediately after the breathing exercises and evaluate the differences between the groups (study and controls). The control group consists of women diagnosed with fibromyalgia who did not participate in breathing sessions. FSFI higher score means better sexual function (maximum score 36).

CONTACTS AND LOCATIONS:
Locations (1):
- Adana City Hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
demographical values could be shared. The questionaries answers are personal so only scale results may be shown.